CLINICAL TRIAL: NCT06695299
Title: Effect of Kinesthetic and Visual Motor Imagery Training on Cervical Position Sense and Balance in Patients With Mechanical Neck Pain
Brief Title: Kinesthetic and Visual Motor Imagery on Cervical Position Sense and Balance in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005399
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Intervention Model Description: the control group which received the selected exercise program and the study group received the same exercise training program in addition to Kinesthetic and Visual Motor Imagery Training
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group received the selected exercise program in addition to Kinesthetic and Visual Motor Imagery Training
  Interventions: Other: selected exercise program; Other: Kinesthetic and Visual Motor Imagery Training
- control group (Experimental): the control group which received the selected exercise program
  Interventions: Other: selected exercise program

INTERVENTIONS:
Other: selected exercise program — therapeutic ultrasound, Static neck exercise, balance exercises
Other: Kinesthetic and Visual Motor Imagery Training — Kinesthetic and Visual Motor Imagery Training During kinesthetic imagery, the participants were asked to feel their body parts without any body motion. During visual imagery, the participants were asked to perform a visual presentation of the motion without any body motion.
  Arms: study group

SUMMARY:
To investigate the Effect of Kinesthetic and Visual Motor Imagery Training on Cervical Position Sense and Balance in Mechanical Neck Pain

DETAILED DESCRIPTION:
Thirty patients with Mechanical Neck Pain will participate in this study. The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to Kinesthetic and Visual Motor Imagery Training, three times per week for four weeks. The evaluation methods are cervical joint position error test, neck disability index, multidirectional reach test and visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* thirty patients with mechanical neck pain,
* Age will range as (35:50) years old
* body mass index (18:29)

Exclusion Criteria:

* difficulty to communicate or to understand program instructions
* any other neurological deficits or orthopaedic abnormalities,
* secondary musculoskeletal complication
* Cervical disc prolapses
* Any other cervical problem
* Spinal stenosis
* Previous spinal surgery

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
cervical joint position error test | four weeks
  The subject will be instructed to perform an active head rotation to one side, after which returns back to the neutral or starting head position.
  The test will be performed in a 3 trials in each direction
Neck disability index | four weeks
  includes 10 items as follows: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation, with a score (0:5) for every point. The maximum score is 50, with the interpretation scoring (no disability = 0: 4, mild disability 5:14, moderate disability 15:24, severe disability 25: 34 and complete disability above 34

SECONDARY OUTCOMES:
Visual analogue scale for pain (VAS-P) | four weeks
  is a method for measuring the intensity of pain on a horizontal straight line of fixed length (10 cm), as the left end of the line showed the greatest pain score & the right end showed the least pain scores, then the patient was asked to put a mark, on the line according to his/her pain sensation, with a higher score representing the higher level of pain
multidirectional reach test | four weeks
  The Multi-Directional Reach Test (MDRT) measures balance and the limits of stability in the anterior-posterior and medial-lateral directions by testing how far an individual can voluntarily reach forward, to the right, to the left, and lean backward, while standing with their feet flat on the ground, shoulder-width apart

CONTACTS AND LOCATIONS:
Locations (1):
- Lama Saad El-Din Mahmoud, Al Jīzah, Select State, Egypt